CLINICAL TRIAL: NCT06059027
Title: Microbes and Respiratory Illnesses, The MARI Study
Brief Title: Microbes and Respiratory Illnesses
Acronym: MARI
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2023-1033; 2U19AI104317 (NIH); Protocol Version 4/30/2025 (Other: UW Madison); A536770 (Other: UW Madison)
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Virus; Asthma
MeSH Terms: conditions — Virus Diseases; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Types of samples collected will include:
  * Blood
  * Nasal Sampling:
  * Nasal Swab: Nasal cells and mucus will be collected by putting a tiny swab (the size of a Q-tip) in the nose moved in and out for 4 seconds. The swab is then removed from the nose. During the baseline visit, the study team will teach the child how to collect this swab at home for the weekly collection. The family will be given the materials to take home to be able to collect the nasal swab at home and mail it back to the study site.
  * Nasal Filter Paper: Nasal secretions will be collected by inserting an absorbent strip into the child's nose for 1-2 minutes.
  * Saliva (spit)
  * Genetic Testing: Some of the tests performed on the child's saliva and nasal samples will be genetic testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TA Cohort: Traditional agrarian (TA) Community Children
- Madison Cohort with Asthma: Madison-area Children with Asthma
- Madison Cohort without Asthma: Madison-area Children without Asthma
- Madison Cohort with Active Respiratory Illness: Madison-area children with active respiratory illness, with or without asthma

SUMMARY:
This study is called the Microbes and Respiratory Illnesses (MARI) Study. Children growing up on farms are exposed to many types of microbes that could be beneficial. It is thought that increased exposure to certain types of microbes early in life helps to develop a healthy immune system and reduce the risk for severe common cold illnesses, breathing problems, and allergies.

DETAILED DESCRIPTION:
Respiratory viruses, most notably rhinoviruses (RV), commonly infect school-age children during the month of September and are a well-known exposure for asthma exacerbations. Allergic sensitization is a risk factor for increased viral respiratory illness burden and wheezing. Nasal Airway Epithelial Cell (NAEC) responses to viral exposure show distinct transcriptional programs that differ in individuals with allergies or asthma. There is a growing body of evidence strongly suggesting nasal airway microbial communities enriched in several commensal bacteria are associated with protection from symptomatic RV infections. Metagenomic sequencing from previously collected nasal samples obtained at age 2 years showed distinct microbial communities and function in the Traditional agrarian (TA) Community Cohort compared to farm and non-farm children. How the early life nasal microbial community can impact risk for viral respiratory infection symptoms and NAEC biology remains an important and unresolved question. To address this important question, this proposal includes an observational study to identify patterns of nasal airway gene expression among three cohorts of school-age children that markedly differ in their susceptibility to respiratory illnesses and wheezing: children from TA/Amish communities, suburban children without asthma, and suburban children with asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or parent guardian must be able to understand and provide informed consent
2. Children ages 4-12 years of age
3. Cohort 1: Family is self-identified as Traditional agrarian (TA) Community member
4. Cohort 2: Madison-area children with parental report of doctor-diagnosed asthma
5. Cohort 3: Madison-area children with no history of asthma by parental report
6. Cohort 4: Madison-area children who have an active respiratory illness

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol
2. Chronic sinusitis (frequent sinus infections)
3. Plans to move out of the area before completing the study
4. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study
5. Enrolled family member

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will be recruited from the LaFarge Medical Clinic and the University of Wisconsin Hospitals and Clinics (Madison area) and the demographics of the participants enrolled will reflect those of the area. It is anticipated that approximately 50% of the study participants will be female. Participation of minority ethnic and racial groups will be encouraged. It is expected that the study population will reflect the demographics of the TA (all White) and Madison (approximately 25% minority) communities. Despite no representation of ethnic minorities, the TA population is a uniquely valuable cohort.
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Respiratory Illness Burden Index (RIBI) | 30 days
  The primary outcome for illness severity will be the Respiratory Illness Burden Index (RIBI), which is calculated as the area under the curve (AUC) for symptom scores and days of illness, as previously described. It is calculated by summing the WURSS (cold symptoms assessment) scores for each day of respiratory illness during the observation period.

SECONDARY OUTCOMES:
Frequency of respiratory illnesses during the monitoring period | 30 days
  Frequency of respiratory illnesses during the monitoring period. Respiratory illnesses are defined as parental perception of respiratory illness symptoms (cold, cough or wheeze) above baseline symptoms.
Virus detection rates in weekly surveillance samples | 30 days
  Virus detection rates in weekly surveillance samples. This will be defined as the detection of a respiratory virus in the weekly nasal mucus specimens.

CONTACTS AND LOCATIONS:
Overall Officials: James Gern, MD, Principal Investigator — UW Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Summary level participant data will be shared but not individual level data.

DOCUMENTS (1):
  • Informed Consent Form (2025-05-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT06059027/ICF_000.pdf